CLINICAL TRIAL: NCT00383487
Title: A Phase II Trial of Calcitriol and Naproxen in Patients With Recurrent Prostate Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Extreme toxicity
Sponsor: Stanford University (Other)
Collaborators: Novacea (Industry)
Responsible Party: Principal Investigator, Sandy Srinivas, Associate Professor of Medicine, Stanford University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PROS0021; 95804 (Other: Stanford University alternate IRB Number)
Record Dates: First submitted 2006-09-29; First posted 2006-10-03 (Estimated); Last update posted 2013-01-28 (Estimated); Status verified 2013-01

CONDITIONS: Prostatic Neoplasms; Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Calcitriol; naproxen-n-butyl nitrate; Naproxen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Calcitriol — 0.5 micrograms/kilogram q weekly
  Other Names: 1,25-Dihydroxycholecalciferol; 1,25-dihydroxyvitamin D3
Drug: Naproxen-n-butyl nitrate — 400 mg BID, oral
  Other Names: Naprosyn

SUMMARY:
To determine whether, in this patient population, treatment with calcitriol and Naproxen is more effective in delaying the growth of prostate cancer than treatment with calcitriol alone as seen in historical controls.

DETAILED DESCRIPTION:
In summary, in vitro and in vivo studies, as well as early phase clinical trial, have shown a promising role for both calcitriol and NSAIDs in the treatment of prostate cancer. Moreover, calcitriol and NSAIDs both exert their antiproliferative effect by decreasing prostaglandin levels, but they do so by different mechanisms. Thus, there is reason to believe that their combined effects on prostaglandins may be synergistic. Preliminary in vitro assays in which calcitriol is given in combination with one of two different NSAIDs (Naprosyn or sulindac) to LNCaP cell lines have indicated such synergy. This observation provides the rational for using them in combination for the treatment of prostate cancer. In addition, it is hoped that any synergy noted would allow for the use of lower doses of NSAIDs.

ELIGIBILITY:
Inclusion Criteria:

* Must give written informed consent
* Histologically confirmed adenocarcinoma of the prostate
* Biochemical relapse after primary radiation therapy or surgery
* Normal testosterone levels
* 3 rising PSA after nadir, with interval between PSA determinations > 2 weeks

Exclusion Criteria:

* Local recurrence by CT scan
* Distant metastases by bone scan
* Hypercalcemia
* Nephrolithiasis
* Renal insufficiency (serum creatinine > 1.8 mg/dl)
* Pancreatitis
* History of ulcer or gastrointestinal bleeding
* More than 6 months of hormone ablation therapy
* Concurrent therapy for prostate cancer
* Uncontrolled HTN
* H/O MI, CVA, TIA
* Known coronary disease/cerebrovascular disease
* Platelet counts <50
* Patients on anticoagulants
* Patients on lithium

Ages: 18 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2005-03; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
PSA response - 50% PSA decline, PSA progression, PSA response duration, progressive disease, time to PSA progression.

SECONDARY OUTCOMES:
Progressive disease in this study's patients, who would be treated with calcitriol and naprosyn, will be compared to that in historical controls of patients treated with calcitriol alone.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Sandy Srinivas, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States